CLINICAL TRIAL: NCT05614024
Title: Neurofeedback During Eating: A Novel Mechanistic Treatment for Bulimia Nervosa
Brief Title: Neurofeedback During Eating for Bulimia Nervosa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Laura Berner, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GCO 21-2078
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Bulimia Nervosa
MeSH Terms: conditions — Bulimia Nervosa

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two conditions, either the experimental or sham neurofeedback arm.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real fNIRS Neurofeedback Arm (Experimental): Participants assigned to the experimental arm will see their true, real-time brain activation (i.e., active real-time neurofeedback) during the neurofeedback session. This activation will be displayed to the participant as a thermometer that will increase as brain activation in the target region increases.
  Interventions: Other: Real fNIRS Neurofeedback
- Sham-Control fNIRS Neurofeedback Arm (Sham Comparator): Participants assigned to the sham-control arm will see false feedback (or a fake signal) that is not connected to their right vlPFC activation during the neurofeedback session.
  Interventions: Other: Sham-Control fNIRS Neurofeedback

INTERVENTIONS:
Other: Real fNIRS Neurofeedback — Participants will be instructed to use real-time fNIRS neurofeedback to non-invasively regulate neural activation associated with symptoms in individuals with bulimia nervosa. During the training, participants will view images on a computer screen, listen to sounds, and consume a shake.
  Arms: Real fNIRS Neurofeedback Arm
Other: Sham-Control fNIRS Neurofeedback — Participants will be instructed to use sham real-time fNIRS neurofeedback to non-invasively regulate neural activation associated with symptoms in individuals with bulimia nervosa. During the training, participants will view images on a computer screen, listen to sounds, and consume a shake.
  Arms: Sham-Control fNIRS Neurofeedback Arm

SUMMARY:
The purpose of this study is to examine the effects of noninvasive prefrontal cortex (PFC) neurofeedback during eating in women with bulimia nervosa (BN) using a wearable brain imaging device, functional near-infrared spectroscopy (fNIRS). The investigators will examine how this training may influence inhibitory control and BN symptoms.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effects of PFC neurofeedback during eating in women with bulimia nervosa (BN) using fNIRS. Specifically, the study aims 1) to demonstrate ventrolateral PFC (vlPFC) neurofeedback target engagement in women with BN using fNIRS; and 2) to link changes in PFC activation to changes in inhibitory control and eating-related symptoms.

Data will be collected from women with BN who will be randomly assigned to one of two group conditions (real or sham-control neurofeedback during eating). Participation includes a phone screening assessment, psychodiagnostic assessment, one in-person evaluation, one neurofeedback session, behavioral tasks, online questionnaires before and after the neurofeedback session, and a remote follow-up assessment.

ELIGIBILITY:
Inclusion criteria:

* Female
* Aged 18 to 45 years
* Meet diagnostic criteria for bulimia nervosa
* Current body mass index greater than or equal to 18.5kg/m2 but under 30kg/m2
* English-speaking

Exclusion criteria:

* Ongoing medical treatment, major medical condition, or psychiatric disorder that may interfere with study variables or participation
* Current psychotherapy focused primarily on eating disorder symptoms
* Pregnancy or planned pregnancy, or lactation during the study period
* Allergy to ingredients in the standardized meal or in the shake

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The prevalence of bulimia nervosa is substantially greater in women than in men. Moreover, prior research suggest that men and women show different neural response patterns during the engagement of inhibitory control, and that satiety differentially impacts the neural function of males and females.
Enrollment: 30 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Functional near-infrared spectroscopy (fNIRS)-measured neural activation and connectivity | approximately 1 hour
  The investigators will evaluate changes in PFC neural activation and connectivity as a function of neurofeedback.
Go/no-go task performance | 2 weeks
  Participants will complete a go/no-go task 1 week before and 1 week after the neurofeedback session to measure inhibitory control.
  Participants behavioral performance on the go/no-go task will be determined by the percentage of incorrect responses made as they are prompted to react to different pictorial stimuli. Participants' percentages of error can range from 0% to 100%. A higher percentage indicates a lower behavioral performance on the task.
Number of loss-of-control eating and purging episodes | 2 weeks
  Frequency of loss-of-control eating and purging episodes. Participants will self-report on how often loss-of-control eating and purging episodes occur using electronic daily diaries in the week before and the week after the neurofeedback session.
Severity of loss-of-control eating scale | 2 weeks
  Severity of loss-of-control eating. Participants will rate the severity of their feelings of control over eating and purging episodes on a Likert-type scale from 0-10. Higher score indicates greater severity of loss of control.

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Berner, Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Center for Computational Psychiatry at the Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: SAP
Time Frame: Immediately following publication and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal to achieve aims in the approved proposal. Proposals should be directed to laura.berner@mssm.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years after article publication via direct request to the investigator.